CLINICAL TRIAL: NCT01057771
Title: Meditation and Exercise for Prevention of Acute Respiratory Infection
Acronym: MEPARI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-0075; R01AT004313 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-27 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Acute Respiratory Infection
Keywords: meditation; exercise; immunity; respiratory infection; influenza; flu shot; immunomodulation
MeSH Terms: conditions — Motor Activity; Respiratory Tract Infections; Influenza, Human | interventions — Meditation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meditation (Experimental): Eight weeks of training in mindfulless meditation. Weekly group sessions of 2.5 hours, with 45 minutes/day of practice.
  Interventions: Behavioral: Meditation
- Exercise (Experimental): Eight weeks of training in moderately strenuous exercise. Weekly group sessions of 2.5 hours, with 45 minutes/day of practice.
  Interventions: Behavioral: Exercise
- Waiting list control (No Intervention): Waiting list control subjects will be treated exactly like those in active intervention groups, but will not receive interventions.

INTERVENTIONS:
Behavioral: Meditation — Eight weeks of training in mindfulless meditation. Weekly group sessions of 2.5 hours, with 45 minutes/day of practice.
  Arms: Meditation
Behavioral: Exercise — Eight weeks of training in moderately strenuous exercise. Weekly group sessions of 2.5 hours, with 45 minutes/day of practice.
  Arms: Exercise

SUMMARY:
The overarching goal of this project is to determine whether mind-body practices such as meditation or exercise can reduce the public health burden of acute respiratory infection. A major secondary goal is to determine whether mindfulness meditation or moderately strenuous exercise can enhance immune processes such as antibody response to influenza vaccination (flu shots). Finally, we want to investigate the influence of stress, optimism, anxiety and positive and negative emotion on immunity and resistance to respiratory infection.

DETAILED DESCRIPTION:
ABSTRACT

Background Preliminary evidence suggests that meditation and exercise may work through interacting psychological and physiological pathways to influence the immune system and reduce infectious respiratory disease.

Methods In this study, women and men aged 50 and older will be randomized to: 1) an 8-week behavioral training program in mindfulness meditation, 2) an intensity, duration and location-matched 8-week exercise training program, or 3) a waiting list control group. Sample size will be N=150 enrolled, with N=50 in each group. The main patient-oriented outcome will be severity-adjusted total days of acute respiratory infection (ARI) illness, as self-reported on the Wisconsin Upper Respiratory Symptom Survey (WURSS-24), a validated questionnaire outcome measure. Nucleic acid based viral identification will verify all symptomatic infections, and the cytokine IL-8 and nasal neutrophil from nasal wash will serve as biomarkers of illness severity. Biomarkers of immune function will include antibody response to influenza immunization (serum IgG, mucosal IgA) and cytokines IFN-γ and IL-10 from cultured ex vivo lymphocytes. Questionnaire measures assessing perceived stress, positive and negative emotion, optimism, and anxiety will be analyzed as potential mediators of immunomodulation and illness prevention.

Timeframe / logistics This will be a 2-year project, with 2 cohorts conducted during a single cold season. The first cohort of N=60 will be randomized and begin interventions in September 2009. The second cohort of N=90 will be randomized and begin interventions in January 2010. Tri-valent influenza vaccination will occur on week 6 of behavioral interventions in both cohorts. Blood for antibody titer and ex vivo cytokine assay will be drawn at baseline, at the end of the 8-week session, and once again 3 months later. Nasal swab for IgA will be done at the same times. Participants will be followed with telephone contact every 2 weeks, with monthly questionnaire instruments, and with daily self-assessments during ARI illness episodes.

Analysis ANOVA-based models will assess effects of meditation and exercise on immune markers and ARI illness. Psychological measures will be assessed as potential mediators of effects of meditation and exercise on ARI illness. Generalized estimating equations, random-effects pattern-mixture models, and hierarchical linear models will be used to assess longitudinal effects, interactions, and covariate mediation.

Section 2. Specific Aims

2.1. Background Acute respiratory infection (ARI) is a leading cause of morbidity and mortality. Influenza is the most pathogenic of the many viruses involved, and hence merits special attention. Protective and ameliorative immune mechanisms are poorly understood, but are associated with various indicators of mental as well as physical health.

A broad literature suggests that regular exercise affects the immune system, positively influences mental health, and protects against ARI illness. A separate and smaller body of evidence suggests that mindfulness meditation may lead to lower stress levels and better mental and physical health. Published evidence from our own study suggests that meditation may enhance antibody (serum IgG) response to influenza vaccination (flu shot) [1].

2.2. Methods & Aims The proposed randomized controlled trial (RCT) will test for effects of meditation and exercise on incidence and severity of ARI illness during an 8-month observation period. Participants (N=150) will be randomized to 1) an 8-week training program in mindfulness meditation, 2)an attention, duration and location-matched program in moderate intensity exercise, or 3) a waiting list control group. Each ARI illness episode will be assessed by a validated questionnaire outcomes instrument, verified with nucleic acid based multiplex viral identification system, and assessed for inflammation with IL-8 assay and neutrophil count from nasal wash. Immunological measures will include antibody response to flu shot (both serum IgG and mucosal IgA) and cytokine indicators of TH1 (IFN-γ) and TH2 (IL-10) immune response, as measured in stimulated ex vivo lymphocyte cell culture. Psychological domains to be assessed include perceived stress, positive and negative emotion, anxiety, and optimism. Immune biomarkers and psychological domains will be assessed as consequences of behavioral interventions, and as predictors of ARI illness. Finally, we will attempt to disentangle the mediating effects of psychological health on immune mechanisms and ARI illness. For example, one hypothesis is that meditation influences the immune system through reduction of stress-related immune dampening mechanisms. That hypothesis would receive support if perceived stress and ARI illness were lowest in the meditation group, and if perceived stress associated more strongly with immune biomarkers and ARI measures than did measures of other psychological domains. We expect that both exercise and meditation will improve psychological health, influence immune biomarkers, and reduce ARI illness burden. However, current evidence is not sufficient to estimate the relative magnitude of these effects, nor to confidently predict whether cellular and/or antibody-mediated immune mechanisms will be implicated.

2.3 Null hypotheses - 2.3.1 Compared to control, an 8-week training program in mindfulness meditation will not lead to statistically significant reductions in number of severity-weighted days of ARI illness. 2.3.2 Compared to control, a matched 8-week exercise training program will not lead to significant reductions in ARI illness. 2.3.3 Meditation training will not enhance either antibody response to flu shot (serum IgG, mucosal IgA), or cytokine expression linked to TH1 and TH2 cell-mediated immune pathways (IFN-γ, IL-10). 2.3.4 Exercise training will not enhance either antibody response to flu shot or cytokine expression from cultured lymphocytes. 2.3.5 Mindfulness meditation training will not lead to improvements in measures of psychological health (perceived stress, positive and negative emotion/affectivity, anxiety, optimism). 2.3.6 Exercise training will not improve these psychological measures. 2.3.7 Immune biomarkers will not predict ARI outcomes. 2.3.8 Psychological measures will not predict ARI outcomes. 2.3.9 The effects of meditation and exercise on psychological measures, immune biomarkers, and ARI illness will not be distinguishable from each other. 2.3.10 Observed effects of meditation and exercise on ARI outcomes will not be explained by either psychological measures or biomarkers of immune mechanisms.

2.4 Justification Influenza and other acute viral infections are responsible for tremendous health burden. Antibody-mediated immunity, responding to vaccination or natural exposure, is only partially effective in conferring protection. Current evidence suggests that cell-mediated immune mechanisms are important in this process. Both antibody-mediated and cell-mediated immune mechanisms have been linked to psychological domains, and appear to decline with aging. Preliminary evidence suggests that both mindfulness meditation and moderate intensity exercise may be at least partially effective in modifying immune response and reducing infectious illness burden. No studies have compared these 2 quite different behavioral intervention techniques. This proposed research would provide new knowledge regarding effects of meditation and exercise training on ARI illness, and immunological and psychological pathways involved.

ELIGIBILITY:
Inclusion Criteria: 1) Aged 50 years or older at study entry. 2) Literacy in English language sufficient for understanding the study protocol and completing questionnaires. 3) Must answer "Yes" to either "Have you had at least 2 colds in the last 12 months?" and/or "On average do you get at least 1 cold per year?" 4) Self-reported ability and willingness to follow through with either exercise or meditation training, or neither, according to randomized allocation. 5) Successful completion of tasks during run-in period, including 2 in-person appointments, 2 phone contacts, and 1 set of homework questionnaires. 6) A score of 14 or lower on the PHQ-9 depression screen, self-reported both at entrance to run-in trial and again just prior to enrollment in the main study. 7) A score of 24 points or higher on the Folstein mini-mental status exam, administered by research personnel at entrance to run-in trial and again just prior to consent and enrollment in the main study.

-

Exclusion Criteria: 1) Physical or medical condition prohibiting adherence to study protocol. Prospective participants must meet the American Heart Association guidelines225 for suitability for an exercise program. Prospective participants will be advised (but not required) to seek their physicians' advice before enrollment. 2) Current or recent use of meditative practice, or previous meditation training. Assessed by answering "Yes" to any of the following questions: Do you meditate on a regular basis? In the last year, have you meditated at least weekly for 2 or more months in a row? Have you ever been trained in meditation? Have you ever been involved in a mindfulness class or mindfulness practice? 3) Potential participants must not engage in moderate exercise more than twice per week or vigorous exercise more than once per week, as assessed by the following questions adapted from the BRFSS classification226 system: On average, how many times per week do you engage in moderate recreational activities such as walking, tennis doubles, ballroom dancing, weight training, or similar activities that last at least 20 minutes per occasion? A) Less than 1 time per week; B) 1 time per week; C) 2 times per week; D) 3 times per week; E) >4 times per week. How many times per week do you engage in vigorous sport and recreational activities such as jogging, swimming, cycling, singles tennis, aerobic dance or other similar activities lasting at least 20 minutes per occasion? A) Less than 1 time per week; B) 1 time per week; C) 2 times per week; D) 3 or more times per week. 4) Immune deficiency or auto-immune disease (eg. HIV/AIDS, lupus, rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease; Co-Investigator Dr. Muller will advise in questionable cases). 5) Current use or forecasted need for immunoactive drugs (eg. steroids, immunosuppressants, chemotherapy); nonsteroidal antiinflammatories will be allowed. 6) Current use or forecasted need for antibiotic or antiviral medications (eg. prophylactic or suppressive therapy for chronic urinary tract infection, recurrent herpes, or other chronic infections. 7) Malignant disease (prospective participants' physicians to advise. Dr. Barrett to make final decision in questionable cases). 8) Function-impairing psychopathology (prospective participants' psychiatrist or psychologist to advise). 9) Influenza vaccination (flu shots) within 6 months prior to enrollment. 10) True egg allergy or true allergic reaction to prior flu shot, either of which would have to include at least one of the following: a) large rash or swelling (more than 12 inches in diameter), b) any swelling in throat, c) any difficulty breathing, d) reaction with hospitalization, or e) anaphylaxis. Reactions that would NOT exclude people: a) local pain or swelling, b) fever, c) malaise, feeling lousy, or d) cold, flu or other infectious illness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Severity-adjusted total days of acute respiratory infection (ARI) illness, as self-reported on the Wisconsin Upper Respiratory Symptom Survey (WURSS-24). Incidence (number) of cold flu episodes and total unadjusted days of illness will also be reported. | 2009-2010 cold season

SECONDARY OUTCOMES:
Immune response to influenza immunization (flu shot): serum IgG, mucosal IgA, and cytokines IFN-γ and IL-10 from cultured ex vivo lymphocytes. Flu shots are given in 6th week of 8 week intervention sessions. | 3 weeks after flu shot
Severity of illness assessed by biomarkers from nasal wash (IL-8, neurophil count) | every cold or flu illness illness episode
Nucleic acid based viral identification will identify pathogen and verify all symptomatic infections | every cold or flu illness episode

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barrett, MD, PhD, Principal Investigator — University of Wisconsin Department of Family Medicine
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Barrett B, Hayney MS, Muller D, Rakel D, Ward A, Obasi CN, Brown R, Zhang Z, Zgierska A, Gern J, West R, Ewers T, Barlow S, Gassman M, Coe CL. Meditation or exercise for preventing acute respiratory infection: a randomized controlled trial. Ann Fam Med. 2012 Jul-Aug;10(4):337-46. doi: 10.1370/afm.1376. PMID 22778122
- [Result] Zgierska A, Obasi CN, Brown R, Ewers T, Muller D, Gassman M, Barlow S, Barrett B. Randomized controlled trial of mindfulness meditation and exercise for the prevention of acute respiratory infection: possible mechanisms of action. Evid Based Complement Alternat Med. 2013;2013:952716. doi: 10.1155/2013/952716. Epub 2013 Sep 29. PMID 24191174
- [Result] Obasi CN, Brown R, Ewers T, Barlow S, Gassman M, Zgierska A, Coe CL, Barrett B. Advantage of meditation over exercise in reducing cold and flu illness is related to improved function and quality of life. Influenza Other Respir Viruses. 2013 Nov;7(6):938-44. doi: 10.1111/irv.12053. Epub 2012 Nov 21. PMID 23170828
- [Result] Hayney MS, Coe CL, Muller D, Obasi CN, Backonja U, Ewers T, Barrett B. Age and psychological influences on immune responses to trivalent inactivated influenza vaccine in the meditation or exercise for preventing acute respiratory infection (MEPARI) trial. Hum Vaccin Immunother. 2014;10(1):83-91. doi: 10.4161/hv.26661. Epub 2013 Oct 7. PMID 24096366
- [Result] Rakel D, Mundt M, Ewers T, Fortney L, Zgierska A, Gassman M, Barrett B. Value associated with mindfulness meditation and moderate exercise intervention in acute respiratory infection: the MEPARI Study. Fam Pract. 2013 Aug;30(4):390-7. doi: 10.1093/fampra/cmt008. Epub 2013 Mar 20. PMID 23515373